CLINICAL TRIAL: NCT01908400
Title: An Open Labeled Clinical Study to Evaluate the Safety and Efficacy of Autologous Bone Marrow Derived Mono Nuclear Stem Cell (BMMNCs) in Patients With Mental Retardation. It is Self Funded (Patients' Own Funding) Clinical Trial
Brief Title: Safety and Efficacy of BMMNCin Patients With Mental Retardation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaitanya Hospital, Pune (Other)
Responsible Party: Principal Investigator, Dr. Sachin Jamadar, Co -investigator, Chaitanya Hospital, Pune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSCC/BMMR/2013//01
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Mental Retardation
Keywords: Mental retardation , stem cell,BMMNC
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BMMNCs (Other): Intravenous transfer of (BMMNCs)
  Interventions: Biological: Intravenous transfer of BMMNC

INTERVENTIONS:
Biological: Intravenous transfer of BMMNC — Intervention therapy , Total 3 doses ,in 30 days ,in 7days interval Intravenous transfer of Autologous Bone Marrow derived Mono Nuclear Stem Cell (BMMNCs)

SUMMARY:
Mental retardation is a condition diagnosed before age 18 that includes below-average general intellectual function, and a lack of the skills necessary for daily living. Mental retardation affects about 1 - 3% of the population. There are many causes of mental retardation, but find a specific reason in only 25% of cases.Bone marrow derived stem cells are used in this condition to prove its safety and efficacy .

ELIGIBILITY:
Inclusion Criteria:

* Age limit: 5 -50
* Primary diagnosis of mental retardation (IQ < 70)
* willingness to undergo Autologous Bone Marrow derived Mono Nuclear Stem Cell (BMMNCs) transplantation.
* To give an informed consent as well as sign the required Informed Consent Form (ICF)/video Consent for the study.
* willingness to regularly visit the hospital / clinic for follow up during the follow up period / on prior agreed time points as per the protocol.

Exclusion Criteria:

* Positive test results for HIV and AIDS complex ,HCV (hepatitis C virus ), HbsAg and Syphilis
* Advanced age that may produce deteriorating cognitive or motor functioning
* Multiple sensory or motor disabilities that will interfere with seeing the stimuli and responding to the computer
* Poor general health

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Binet-Kamat Test | 1 YEAR
  CHANGE in IQ as measured by Binet-Kamat Test

SECONDARY OUTCOMES:
Vineland Social Maturity Scale | baseline and 12 months
  CHANGE in Social Quotient as measured by Vineland Social Maturity Scale

CONTACTS AND LOCATIONS:
Overall Officials: ANANT E BAGUL, MS ORTHO, Principal Investigator — Chaitanya Hospital
Locations (1):
- Chaitanya Hospital, Pune, Maharashtra, India